CLINICAL TRIAL: NCT01941290
Title: Biotronik-Safety and Performance Registry for an All-comers Diabetic Patient Population With the Limus Eluting Orsiro Stent System Within Daily Clinical Practice-III Asia
Brief Title: BIOFLOW III Asia Registry Orsiro Stent System
Status: Completed | Type: Observational
Sponsor: BIOTRONIK Asia Pacific Pte Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: G1206
Record Dates: First submitted 2013-09-03; First posted 2013-09-13 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Diabetes Mellitus Type 1 or 2
Keywords: International; Multicenter; Observational registry; Orsiro Drug Eluting Stents (DES); Stenting; Treatment of Coronary Artery Disease; Coronary Revascularization; Percutaneous Coronary Intervention (PCI); Diabetes Mellitus Type 1; Diabetes Mellitus Type 2; STEMI; NSTEMI; Ischemia; Angina; Subgroups; Acute Myocardial Infarction; Small Vessels; Chronic Total Occlusion
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Ischemia; Angina Pectoris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Orsiro

SUMMARY:
Cliflical evaluation of th' Orsiro LESS 10 diabetic subjects requiring coronary revasculariza t ion with Drug Eluting Stefl ts (DES) .880 subjects will be enrolled in this registry. The sample subjects size may be increased in order to reach the subgroup sizes (Small Vessel and AMI).

DETAILED DESCRIPTION:
For the majority of Coronary Artery Disease (CAD), treatment with Percutaneous Transluminal Coronary Angioplasty (PTCA) provides high initial procedural success. However, the medium to long-term complications range from rather immediate elastic recoil or vessel contraction to longer processes like smooth muscle cell proliferation and excessive production of extra cellular matrix, thrombus formation and atherosclerotic changes like restenosis or angiographic re-narrowing. The reported incidence of restenosis after PTCA ranges from 30%-50%. Such rates of recurrence have serious economic consequences. Bare Metal Stents (BMS), designed to address the limitations of PTCA, reduced the angiographic and clinical restenosis rates in de novo lesions compared to PTCA alone and decreased the need for CABG. BMS substantially reduced the incidence of abrupt artery closure, but restenosis still occurred in about 20%-40% of cases, necessitating repeat procedures. The invention of Drug Eluting Stents (DES) significantly improved on the principle of BMS by adding an antiproliferative drug (directly immobilized on the stent surface or released from a polymer matrix), which inhibits neointimal hyperplasia. The introduction of DES greatly reduced the incidence of restenosis and resulted in a better safety profile as compared to BMS with systemic drug administration. These advantages and a lower cost compared to surgical interventions has made DES an attractive option to treat coronary artery disease.

An interesting group of analysis resulted to be diabetic patients. It has been concluded that the incidence of both nonocclusive and occlusive restenosis is higher in diabetic subjects after stenting as judged from comparison with historical control subjects. Results implicate accelerated restenosis as both a consequence of diabetes and a cause for increased mortality after PCI in diabetic patient.

Therefore this observational registry has been designed for the clinical evaluation of the Orsiro LESS in diabetic subjects (Diabetic patients type 1 or 2) requiring coronary revascularization with Drug Eluting Stents (DES). Results will contribute to the collection of clinical evidence for the clinical performance and safety of the Orsiro Drug Eluting Stent System in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria
* Diabetes Mellitus:

  * Known Diabetic on Pharmacological treatment.
  * ACS NSTEMI with documented Hb A1c> 7%, even if not on Pharmacological treatment for diabetes.
* Patient has Symptomatic coronary artery disease
* Target lesion must be a de novo lesion located in a native coronary artery with reference vessel diameter ≥2.25 mm & ≤4.00 mm, lesion length ≤40 mm by visual estimate
* Patient should be receiving up to 3 stents and up to 2 stents per artery.
* Target lesion must be in a major coronary artery or branch with visually estimated stenosis ≥50% & <100% with TIMI flow≥1.
* Subject provides signed informed consent for data release
* Subject is geographically stable and willing to comply with protocol required follow ups
* Subject is ≥ 18 years of age

Exclusion Criteria:

* Pregnant and/or breast-feeding females who intend to become pregnant during the period of the registry
* Untreatable intolerance to aspirin, clopidogrel, ticlopidine, heparin or any other anticoagulation / antiplatelet therapy required for PCI, stainless steel, Sirolimus or contrast media
* Planned surgery within 6 months of PCI unless dual antiplatelet therapy will be maintained
* Currently participating in another study and primary endpoint is not reached yet
* If the subject has a high probability that a procedure other than predilatation, stent implantation and post dilatation will be required at time of index procedure for treatment of target vessel (e.g. atherectomy, cutting balloon or brachytherapy).
* Patients admitted for treatment of Diabetic ketoacidosis ≥ 2 times in the past Six months (Brittle Diabetics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic Subjects requiring coronary revascularization with Drug eluting Stent (DES)
Sampling Method: Non-Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  Composite of cardiac death, target vessel Q-wave or non Q-wave Myocardial Infarction (MI), Emergent Coronary Artery Bypass Graft (CABG), clinically driven Target Lesion Revascularization (TLR)

SECONDARY OUTCOMES:
Target Lesion Failure (TLF) | 6 months
  Composite of cardiac death, target vessel Q-wave or non Q-wave Myocardial Infarction (MI), Emergent Coronary Artery Bypass Graft (CABG), clinically driven Target Lesion Revascularization (TLR)
Clinically Driven Target Vessel Revascularization (TVR) | 6 and 12 months
  Any repeat revascularization of the target vessel.
Clinically Driven Target Lesion Revascularization (TLR) | 6 and 12 months
  Any repeat revascularization of the target lestion.
Stent Thrombosis rate using ARC definition | 12 months
  Definite, Probable and Possible Stent ThrombOsis
Clinical device success | Participants will be followed for the duration of hospital stay, an expected average of 2 days
  Successful delivery and deployment of the investigational stent(s) at the intended target lesion and successful withdrawal of the stent delivery system with attainment of a final residual stenosis of less than 50% by visual estimation and without use of a device outside the assigned treatment strategy.
Clinical Procedure Success | Participants will be followed for the duration of hospital stay, an expected average of 2 days
  Successful delivery and deployment of the investigational stent(s) at the intended target lesion and successful withdrawal of the stent delivery system with attainment of a final residual stenosis of less than 50% of the target lesion as observed by visual estimate without using any adjunctive device* without the occurrence of ischemia-driven major adverse cardiac event (ID-MACE) during the hospital stay to a maximum of the first seven days post index procedure.
  In case of multiple lesions treatment, all treated lesions must meet the clinical procedural success.
  * Apart from post-dilatation with a non-compliant balloon

CONTACTS AND LOCATIONS:
Overall Officials: Upendra Kaul, Dr, Principal Investigator — Fortis Escorts Heart Institute
Locations (19):
- Queen Mary Hospital, Hong Kong, China
- India (12):
  - KMC Manjpal, Manial, Karnataka
  - Fortis Hospitals-Bannerghatta Road, Bangalore
  - Fortis Hospitals Bannerghatta Road, Bangalore
  - GKNM Hospital, Coimbatore
  - Divine Heart and Multi-Specialty Hospital, Lucknow
  - King George Medical University, Lucknow
  - Fortis Hospital, Mohali
  - Holy Family Hospital, Mumbai
  - BLK Super Speciality Hospital, New Delhi
  - Dharma Vira Heart Centre, Sir Ganga Ram Hospital, New Delhi
  - Fortis Escort Heart Institute, New Delhi
  - Ruby Hall Clinic, Pune
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- Sri Lanka (3):
  - Lanka Hospital, Colombo
  - National Hospital of Sri Lanka, Colombo
  - Sri Jaiewardenepura General Hospital, Colombo
- Vietnam (2):
  - Bach Mai Hospital, Hanoi
  - Cho Ray Hospital, Ho Chi Minh City